CLINICAL TRIAL: NCT00959491
Title: A Prospective Study of a New Immunological Fecal Occult Blood Test in Patients Referred for Colonoscopy
Brief Title: A Prospective Study of a New Immunological Fecal Occult Blood Test
Acronym: RLHV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Gastroenterology, Cuba (Other)
Responsible Party: Luis Calzadilla Bertot, National Institute of Gastroenterology
Other Study IDs: RH-9
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Colonoscopy; Occult Blood; Immunologic Tests
Keywords: Colonoscopy; Occult Blood; Fecal

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One fecal sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colonoscopy indication: All outpatients referred to colonoscopy according to inclusion criteria in the specified period time of one year .

SUMMARY:
The purpose of the investigators study is to evaluate the diagnostic ability of a new immunological fecal occult blood test in Cuban patients undergoing colonoscopy .

DETAILED DESCRIPTION:
Colorectal cancer is a major cause of cancer deaths in many countries. Therefore, the importance of screening for the early detection of colorectal cancer is evident. Fecal occult blood screening is proving to be an effective tool for detecting premalignant adenomas and colon cancer since the guaiac-based test was introduced in the late 1960s. However, several immunochemical fecal occult blood tests (IFOBTs) have become commercially available and the majority of these have demonstrated equal or superior sensitivities and specificities than the guaiac-based tests. Therefore, IFOBTs are replacing guaiac based tests despite their higher costs.In this study we evaluate the diagnostic accuracy of a new IFOBT and compare with the findings on colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients (men or women) that are >18 years of age referred to colonoscopy.

Exclusion Criteria:

* Visible rectal bleeding
* Known diagnosis of inflammatory bowel disease
* Hematuria
* Menstruation at the time of obtaining a stool specimen
* Patients taking medication such as non steroids anti inflammatory drugs and anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Havana City admitted at the investigation center.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Luis C Bertot, MD, Principal Investigator — National Institute of Gastroenterology , Havana, Cuba
Locations (1):
- National Institute of Gastroenterology, Havana, La Habana, Cuba